CLINICAL TRIAL: NCT01097850
Title: Prospective Randomized Controlled Open-label Trial of a Topical Henna Preparation for the Treatment of Hand-Foot Skin Syndrome and Its Associated Symptoms
Brief Title: Topical Henna Preparation for the Treatment of Hand Foot Skin Syndrome
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No subject accrual.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Dennis West, Professor in Dermatology and Pediatrics, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 09D1
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Hand Foot Skin Syndrome
Keywords: hand foot skin syndrome; palmar plantar erythrodysesthesia; doxorubicin; capecitabine
MeSH Terms: conditions — Hand-Foot Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right (Other): Application of henna paste to right hand/foot plus CeraVe moisturizer
  Interventions: Drug: henna paste
- Left (Other): Application of henna paste to the left hand/foot plus CeraVe moisturizer
  Interventions: Drug: henna paste

INTERVENTIONS:
Drug: henna paste — Henna paste will be applied to either the left hand/foot or right hand/foot, along with CeraVe moisturizer to both hands/feet

SUMMARY:
The purpose of this study is to determine whether henna paste is effective in the treatment of hand-foot skin syndrome, induced by the drugs Capecitabine and pegylated liposomal doxorubicin.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving capecitabine and/or pegylated liposomal doxorubicin as monotherapy or in combination with other agents
* New diagnosis of active hand-foot skin reaction (on bilateral hands and/or bilateral feet) of 1-3 toxicity as defined by the NCI-CTCAE version 4.0 grading scale with onset of symptoms within the last thirty days
* Patients must be 18 years or older
* Patients must provide written informed consent to participate in the study

Exclusion Criteria:

* Patients with pre-existing dermatological condition affecting the hands or feet that may limit the interpretation of results
* Known allergy to natural henna
* Patients with a previous history of HFS
* History of G6PD deficiency as determined by screening bloodwork

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
• To compare the severity of HFS in subjects receiving topical natural henna paste treatment along with using CeraVe™ moisturizing cream concurrently on the treatment side and using only CeraVe™ moisturizing cream on the control side. | 3 weeks

SECONDARY OUTCOMES:
To examine quality of life, comparing natural henna treatment versus CeraVe™ alone, using the Skindex-16 questionnaire | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lio, MD, Principal Investigator — Northwestern University